CLINICAL TRIAL: NCT04428359
Title: A Comparative Study to Assess Efficacy of Intralesional MMR (Measles, Mumps, Rubella) Vaccine and Intralesional Vitamin D3 in Treatment of Warts
Brief Title: A Comparative Study to Assess Efficacy of Intralesional MMR Vaccine and Intralesional Vitamin D3 in Treatment of Warts
Acronym: MMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Bibisha Baaniya, Junior Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRC/1607/019; 858 - 2019 (Other: Nepal Health Research Council)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Verruca Viral
Keywords: Warts; Intralesional; MMR; Vitamin D; Immunotherapy
MeSH Terms: conditions — Warts | interventions — Measles-Mumps-Rubella Vaccine; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Group A - will receive IL MMR Group B- will receive IL Vitamin D3
Who Masked: Participant
Masking Description: Only patients will be blinded to the randomization and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measles, Mumps, Rubella vaccine (Experimental): All Group A patients will receive intralesional MMR.
  Interventions: Drug: Measles-Mumps-Rubella Vaccine
- Vitamin D3 (Experimental): All Group B patients will receive intralesional Vitamin D3
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Measles-Mumps-Rubella Vaccine — Group A patients will receive intralesional injection of upto 0.5 mL of reconstituted MMR vaccine into a single or a maximum of 5 warts at a time in case of multiple warts. Intralesional injection will be given every three weeks for a maximum of 5 doses or until complete resolution, whichever is earlier.
  Other Names: MMR
  Arms: Measles, Mumps, Rubella vaccine
Drug: Vit D — Group B patients will receive a maximum of 0.5 mL Inj. Vitamin D3 (600,000 IU; 15mg/ml) in each session after injection of IL lignocaine with 31 G insulin syringe. In cases of multiple warts, a maximum of 5 warts will be injected at a time. The session will be done at 3 weekly intervals for a maximum of 5 sessions or until complete resolution of warts, whichever is earlier
  Other Names: Vitamin D3
  Arms: Vitamin D3

SUMMARY:
Common warts are papulonodular epidermal lesions caused by human papillomavirus (HPV) usually by the strains 1, 2, 4, 27 or 57. Cutaneous warts occur in 7% to 10% of the general population, with a maximum incidence between 12 and 16 years. There are multiple destructive treatment modalities of wart but they have many adverse effects. Hence immunotherapy is becoming popular in treatment of warts. It is believed that the injection to the HPV-infected tissue induces a strong nonspecific pro-inflammatory signal and attracts the antigen-presenting cells. Which then promotes a Th1 cytokine response and leads to delayed-type hypersensitivity reaction leading to the eradication of the HPV-infected cells.

We are undertaking a study to evaluate and compare the safety and efficacy of 2 such immunotherapeutic agents namely, IL measles, mumps and rubella (MMR) vaccine versus IL vitamin D3 for the treatment of warts.

RESEARCH HYPOTHESIS Null Hypotheses: IL MMR vaccine is not better than IL Vitamin D in the treatment of wart Alternative hypothesis: IL MMR vaccine is better than IL Vitamin D in the treatment of wart

Method: A total of 60 patients will be included in the study, 30 in each group. Group A and Group B patients will be injected with 0.5 ml of IL MMR and 0.5 ml of IL vitamin D3 respectively into a single or a maximum of 5 warts at a time in case of multiple warts. The IL injection will be given every 3 weeks for a maximum of 5 doses. Clinical assessment will be done by taking photographs and measurements at baseline, before each treatment session, and 3 months after the completion of treatment. The response will be evaluated by a decrease in the size and number of the wart(s) and photographic comparison. The response will be considered complete if there is a complete clearance of the wart(s), good if the wart(s) will regress in size by 75-99%, moderate if they regress by 50-74% and no or mild if there will be a 0-49% decrease in wart(s). Immediate and late side effects of MMR and Vitamin D will be evaluated after each session. Follow up will be made monthly for 3 months to detect any recurrence. Quality of life (QoL) will be measured in wart patients, using the Nepali version of the dermatology life quality index (DLQI) questionnaire before initiation of treatment and at the end of follow up.

Statistical analysis will be done using Statistical Package for the Social Sciences 10.5 version.

DETAILED DESCRIPTION:
INTRODUCTION Warts are common skin conditions resulting from infection of keratinocytes by human papillomavirus (HPV). After infection of the basal layer, there is clonal proliferation leading to epidermal thickening and hyperkeratinization and eventually results in a visible wart. HPVs are ubiquitous, epitheliotropic non-enveloped small double-stranded DNA viruses. Over 150 types of HPVs have been identified. Among them verruca vulgaris are usually caused by HPV types 1, 2, 4, 27 or 57, and plane warts by HPV types 3 or 10.

Cutaneous warts occur in 7% to 10% of the general population, with a maximum incidence between the ages of 12 and 16 years. In children, clearance can occur after only a few months, with 50% at 1 year and about 65%-78% by 2 years. The rate of clearance is influenced by factors like virus strain, host immune status, extent and duration of warts. The transmission of warts occurs from direct contact or indirectly via fomites.

There are multiple destructive, antiproliferative and antiviral agents in treatment of warts. Other modalities include hypnotherapy, acupuncture, local hyperthermia, therapeutic vaccination and combinations of the previous agents. Destructive therapies usually come with many adverse effects hence immunotherapy is becoming more popular, especially in the treatment of refractory cutaneous and genital warts. These include various topical, intralesional (IL) and systemic agents. IL Measles, Mumps, rubella (MMR) and IL vitamin D3 are examples of immunotherapeutic agents.

Immunotherapy is defined as a type of biological therapy that uses substances to stimulate or suppress the immune system to help the body fight cancer, infection, and other diseases. Immunotherapy can affect the immune system in general or can be cell-specific.

Immunotherapy is believed to induce a strong nonspecific pro-inflammatory signal and attract the antigen-presenting cells. This is associated with the release of cytokines such as IL-2, IL-8, IL-12, IL-I8, tumor necrosis factor-α, and interferon-γ. This then promotes a Th1 cytokine response which leads to the activation of delayed-type hypersensitivity reaction leading to the eradication of the HPV-infected cells. Furthermore, the trauma of the injection may also cause a resolution in previously sensitized individuals. Vitamin D3 is also claimed to regulate epidermal cell differentiation and proliferation and may modulate cytokine production through its action upon vitamin D receptors (VDRs). Since IL antigen immunotherapy enhances recognition of the virus by the immune system it causes clearance of both treated and untreated lesions and helps to prevent future clinical infection through induction of long-term acquired immunity to HPV.

MMR vaccine is included in immunization schedule of Nepal so pre-sensitization skin test is not needed as all patients are expected to be immune. The presence of 3 different antigens in MMR increases the sensitivity to the injected antigen and decreases the likelihood of anergy. Side effects of MMR include pain during injection, flu-like symptoms, pruritus and burning sensation.

IL vitamin D is a novel addition to therapies in warts as it is a simple, effective, well-tolerable, and inexpensive method with negligible local and systemic side effects. Side effects of Vitamin D3 include transient mild to moderate pain, edema at the site of injection and mild erythema. Additionally, it would be safer to monitor serum vitamin D and calcium levels before and after intralesional vitamin D treatment to prevent possible hypervitaminosis D.

RATIONALE Intralesional Immunotherapy is an emerging method of treatment of wart in which injection in a single wart causes the resolution of distant warts as well. Compared to other destructive modalities, it is more effective and comfortable for the patient as it obviates the need for individual treatment of each wart. In addition it has a lower rate of recurrence, avoids adverse effects such as scarring, is more cost-effective in multiple warts and decreases the time a physician has to spend on each patient. Further both injection MMR and Vitamin D3 are readily available as compared to other immunotherapeutic agents like purified protein derivative and candida antigen.

IL MMR vaccine has been used for a longer time than IL vitamin D and there are more comparative studies showing efficacy of MMR vaccine with rates of clearance ranging from 70.4% to 82.4%. The clearance rates for IL vitamin D ranges from 40% to 90%.

The advantages of vitamin D over MMR vaccine are cost-effectiveness, non-requirement of maintenance of cold chain, easy availability, and feasibility of use in immunosuppressed patients.

As per Institute of Medicine (IOM), the tolerable upper intake of vitamin D is 4000 IU/day for anyone older than 9 years such that annual maximum dose will be 1,460,000 IU. The total amount of vitamin D that we will be administering will be 1,500,000 IU. Furthermore, since we are giving it intralesionally systemic absorption is likely to be low although data on exact amount of IL vitamin D that gets absorbed systemically is not available. In other studies, patients have been evaluated clinically for signs and symptoms of hypervitaminosis D however, no signs of toxicity were observed.

As per our literature search,

1. No previous studies on immunotherapy in wart have been conducted in our country
2. No comparative studies have been done to compare IL MMR and IL vitamin D3 in treatment of wart hence we aim to establish efficacy of each and compare the two.

OBJECTIVES

Primary Objectives:

1. To determine the efficacy of IL MMR vaccine in the treatment of Wart
2. To determine the efficacy of IL vitamin D in the treatment of wart
3. To compare the efficacy of IL MMR vaccine and IL Vitamin D

Secondary Objective:

1. To determine the clinical and demographic profile of patients with different types of warts visiting Dermatology outpatient department(OPD) of BP Koirala Institute of Health Sciences (BPKIHS)
2. To determine the side effects of IL MMR vaccine and IL Vitamin D in treatment of wart
3. To determine Dermatology life quality index (DLQI) in wart patients.

Operational definition Wart - clinical diagnosis made by a dermatologist Complete response (100%)- Complete disappearance of warts including distant ones and skin texture at the site is restored to normal Excellent response (75-99%)-Reduction in size and number including distant ones and few residual warts still visible Good response (50-74%)-Some reduction in size only including that of distant ones but no decrease in number of warts Poor or no response (0-49%)-No significant change in size and number of warts Recurrence- Recurrence during the study period

MATERIALS AND METHODOLOGY Materials: Study population will be all patients clinically diagnosed with warts visiting the Dermatology OPD of BPKIHS, Dharan.

Study design: Prospective comparative longitudinal study Study Period: Probable duration of the study will be 1 year after approval from the Institutional Review Committee (IRC) and Nepal Health Research Council (NHRC) Ethical Clearance: Taken from IRC, BPKIHS and NHRC Conflict of interest: None Sampling Technique: Census method with all consecutive patients meeting inclusion criteria for initial 6 months Sample size The study considers a 95% confidence interval, 80% power to estimate sample size. According to the literature review, it was found that there was 84.6% and 40% improvement in MMR and Vitamin D respectively.

Now using the sample size estimation formula for 2 proportion {(Zα√2p(1-p)+ Z1-β√((p1(1-p1) p2(1-p2)}2))/(p1-p2)2 Where n= sample size for each group p1 = 0.846 p2 = 0.40 p= (p1 +p2)/2 Zα=1.96 Z1-β = 1.28 Using above formula, n= 12.3 The formula for actual sample size is n/4{1+√(1+4/n|p1-p2|)}2 na = 16.48 Adding 10% in calculated value to reduce bias sampling technique, the minimum sample size in each group is 18.13 =19 Considering loss of follow up, sample size in each group= 30 Total sample size= 60

Methodology Based on the computer generated random number table, patients satisfying inclusion criteria will be assigned to either Group A or Group B once they come to OPD. Informed consent will be taken and detailed information including personal data, past history, medical history, drug history, clinical data like site, size, number and distribution of lesions will be recorded in preset pro forma. Photographs of the lesions will be taken before the first treatment session, in every treatment session and 3 months after last session.

Group A Freeze-dried MMR vaccine single-use vials stored at 2°C-8°C will be reconstituted with 0.5 mL of distilled water immediately before IL use. If reconstituted vaccine is not used within 8 hours it must be discarded. All Group A patients will receive IL injection of upto 0.5 mL of reconstituted MMR vaccine into a single or a maximum of 5 warts at a time in case of multiple warts with 31 G insulin syringe with beveled edge facing upward. Amount of injection on each wart will depend on the size of each wart. The injection will be given every three weeks for a maximum of 5 doses.

Group B All Group B patients will receive a maximum of 0.5 mL Inj. Vitamin D3 (600,000 IU; 15mg/ml) in each session after injection of IL lignocaine with 31 G insulin syringe. In cases of multiple warts, a maximum of 5 warts will be injected at a time. Amount of injection on each wart will depend on the size of each wart. The session will be done at 3 weekly intervals for a maximum of 5 sessions or until complete resolution of warts, whichever is earlier. In patients of group B serum vitamin D level will be measured after 20 days of 3rd dose and 1 month after the last dose to ensure safe monitoring.

Patient and physician global assessment using 'Visual Analog Scale score' and photographic comparison will be used to assess the response to treatment as mentioned in operational definition. Immediate and late adverse effects in both groups will be evaluated after each treatment session. Necessary investigations and intervention will be done if needed. Follow up will be made monthly for 3 months to detect any recurrence.

Quality of Life(QoL) QoL will be measured in wart patients, using the Nepali version of the dermatology life quality index (DLQI) questionnaire before initiation of treatment and at the end of follow up. DLQI contains 10 questions that involves 6 sections: symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Questions 1 and 2 assess symptoms and feelings; 3 and 4, daily activities; 5 and 6, leisure; 7, work and school; 8 and 9, personal relationships and 10, treatment. The clinically meaningful change or reduction in the DLQI score is measured as the change in score from one band to the other.

Statistical analysis

1. Data handling: Data will be entered in Microsoft Excel 2010 and statistical analysis will be done using Statistical Package for the Social Sciences 10.5 version
2. Coding: Alpha numerical code will be used
3. Monitoring: Data will be entered after every day of work and supervised by guide.
4. Statistical Analysis:

   1. Chi square test to compare the categorical data between the groups.
   2. Paired t test for comparing normally distributed continuous variables at different time point within the group
   3. Independent 't' test for comparing normally distributed continuous variables at different time point between the groups
   4. Wilcoxon signed rank test to compare the not normally distributed variables, ordinal data
   5. Mann- Whitney U test to compare the not normally distributed variables, ordinal data.
   6. Kaplan-Meier curves to compare the response rate on each follow up visit between the groups.

Test of significance will be considered when value of p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed patients who have more than three warts or single wart in difficult to treat sites (periungual, palms and soles)

Exclusion Criteria:

1. Patients not under any systemic or topical treatment of warts for the last four weeks
2. Patients with a past history of an allergic response to MMR or any other vaccine or Vitamin D
3. Patients with current acute febrile illness or any bacterial infection
4. Immunosuppressed patients
5. Pregnant or lactating women
6. Patients having a past history of asthma, allergic skin disorders or convulsions
7. Patients with keloidal tendency
8. Patient refusal for consent
9. Treating physician's decision to give other treatment modality
10. Patients with hypervitaminosis D, muscle weakness, bone pain, altered sensorium

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bibisha Baaniya, MBBS, Principal Investigator — B.P. Koirala Institute of Health Sciences
Locations (1):
- BP Koirala Institute of Health Sciences, Dharān, One, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilkenny M, Marks R. The descriptive epidemiology of warts in the community. Australas J Dermatol. 1996 May;37(2):80-6. doi: 10.1111/j.1440-0960.1996.tb01010.x. PMID 8687332
- [Background] Sterling JC, Gibbs S, Haque Hussain SS, Mohd Mustapa MF, Handfield-Jones SE. British Association of Dermatologists' guidelines for the management of cutaneous warts 2014. Br J Dermatol. 2014 Oct;171(4):696-712. doi: 10.1111/bjd.13310. Epub 2014 Oct 1. No abstract available. PMID 25273231
- [Background] Bruggink SC, Eekhof JA, Egberts PF, van Blijswijk SC, Assendelft WJ, Gussekloo J. Natural course of cutaneous warts among primary schoolchildren: a prospective cohort study. Ann Fam Med. 2013 Sep-Oct;11(5):437-41. doi: 10.1370/afm.1508. PMID 24019275
- [Background] DaCruz DJ. Guidelines for management of asthma. BMJ. 1990 Dec 1;301(6763):1276-7. doi: 10.1136/bmj.301.6763.1276-c. No abstract available. PMID 2271835
- [Background] Lipke MM. An armamentarium of wart treatments. Clin Med Res. 2006 Dec;4(4):273-93. doi: 10.3121/cmr.4.4.273. PMID 17210977
- [Background] Leung L. Recalcitrant nongenital warts. Aust Fam Physician. 2011 Jan-Feb;40(1-2):40-2. PMID 21301692
- [Background] Goihman-Yahr M, Goldblum OM. Immunotherapy and warts: a point of view. Clin Dermatol. 2008 Mar-Apr;26(2):223-5. doi: 10.1016/j.clindermatol.2007.10.011. No abstract available. PMID 18472063
- [Background] Bacelieri R, Johnson SM. Cutaneous warts: an evidence-based approach to therapy. Am Fam Physician. 2005 Aug 15;72(4):647-52. PMID 16127954
- [Background] Khanal S, Sedai TR, Choudary GR, Giri JN, Bohara R, Pant R, Gautam M, Sharapov UM, Goodson JL, Alexander J, Dabbagh A, Strebel P, Perry RT, Bah S, Abeysinghe N, Thapa A. Progress Toward Measles Elimination - Nepal, 2007-2014. MMWR Morb Mortal Wkly Rep. 2016 Mar 4;65(8):206-10. doi: 10.15585/mmwr.mm6508a3. PMID 26937619
- [Background] Liu PT, Stenger S, Li H, Wenzel L, Tan BH, Krutzik SR, Ochoa MT, Schauber J, Wu K, Meinken C, Kamen DL, Wagner M, Bals R, Steinmeyer A, Zugel U, Gallo RL, Eisenberg D, Hewison M, Hollis BW, Adams JS, Bloom BR, Modlin RL. Toll-like receptor triggering of a vitamin D-mediated human antimicrobial response. Science. 2006 Mar 24;311(5768):1770-3. doi: 10.1126/science.1123933. Epub 2006 Feb 23. PMID 16497887
- [Background] Silverberg JI, Silverberg NB. The U.S. prevalence of common warts in childhood: a population-based study. J Invest Dermatol. 2013 Dec;133(12):2788-2790. doi: 10.1038/jid.2013.226. Epub 2013 May 8. No abstract available. PMID 23657500
- [Background] Liu J, Li H, Yang F, Ren Y, Xia T, Zhao Z, Cao X, Wang Z, Yin M, Lu S. Epidemiology and Clinical Profile of Cutaneous Warts in Chinese College Students: A Cross-Sectional and Follow-Up Study. Sci Rep. 2018 Oct 18;8(1):15450. doi: 10.1038/s41598-018-33511-x. PMID 30337549
- [Background] Laurent R, Kienzler JL. Epidemiology of HPV infections. Clin Dermatol. 1985 Oct-Dec;3(4):64-70. doi: 10.1016/0738-081x(85)90050-1. No abstract available. PMID 3880029
- [Background] Jablonska S, Orth G, Obalek S, Croissant O. Cutaneous warts. Clinical, histologic, and virologic correlations. Clin Dermatol. 1985 Oct-Dec;3(4):71-82. doi: 10.1016/0738-081x(85)90051-3. No abstract available. PMID 2850861
- [Result] Dhope A, Madke B, Singh AL. Effect of Measles Mumps Rubella Vaccine in Treatment of Common Warts. 2018;(2):81-84. doi:10.4103/ijdd.ijdd
- [Result] Salman S, Ahmed MS, Ibrahim AM, Mattar OM, El-Shirbiny H, Sarsik S, Afifi AM, Anis RM, Yakoub Agha NA, Abushouk AI. Intralesional immunotherapy for the treatment of warts: A network meta-analysis. J Am Acad Dermatol. 2019 Apr;80(4):922-930.e4. doi: 10.1016/j.jaad.2018.07.003. Epub 2018 Jul 10. PMID 30003983
- [Result] Nofal A, Nofal E, Yosef A, Nofal H. Treatment of recalcitrant warts with intralesional measles, mumps, and rubella vaccine: a promising approach. Int J Dermatol. 2015 Jun;54(6):667-71. doi: 10.1111/ijd.12480. Epub 2014 Jul 29. PMID 25070525
- [Result] Thappa DM, Chiramel MJ. Evolving role of immunotherapy in the treatment of refractory warts. Indian Dermatol Online J. 2016 Sep-Oct;7(5):364-370. doi: 10.4103/2229-5178.190487. PMID 27730031
- [Result] Kareem IMA, Ibrahim IM, Mohammed SFF, Ahmed AA. Effectiveness of intralesional vitamin D3 injection in the treatment of common warts: Single-blinded placebo-controlled study. Dermatol Ther. 2019 May;32(3):e12882. doi: 10.1111/dth.12882. Epub 2019 Apr 16. PMID 30920098
- [Result] Nofal A, Salah E, Nofal E, Yosef A. Intralesional antigen immunotherapy for the treatment of warts: current concepts and future prospects. Am J Clin Dermatol. 2013 Aug;14(4):253-60. doi: 10.1007/s40257-013-0018-8. PMID 23813361
- [Result] Abd-Elazeim FM, Mohammed GF, Fathy A, Mohamed RW. Evaluation of IL-12 serum level in patients with recalcitrant multiple common warts, treated by intralesional tuberculin antigen. J Dermatolog Treat. 2014 Jun;25(3):264-7. doi: 10.3109/09546634.2013.768760. Epub 2013 May 6. PMID 23336207
- [Result] Horn TD, Johnson SM, Helm RM, Roberson PK. Intralesional immunotherapy of warts with mumps, Candida, and Trichophyton skin test antigens: a single-blinded, randomized, and controlled trial. Arch Dermatol. 2005 May;141(5):589-94. doi: 10.1001/archderm.141.5.589. PMID 15897380
- [Result] Kus S, Ergun T, Gun D, Akin O. Intralesional tuberculin for treatment of refractory warts. J Eur Acad Dermatol Venereol. 2005 Jul;19(4):515-6. doi: 10.1111/j.1468-3083.2004.01176.x. No abstract available. PMID 15987315
- [Result] Na CH, Choi H, Song SH, Kim MS, Shin BS. Two-year experience of using the measles, mumps and rubella vaccine as intralesional immunotherapy for warts. Clin Exp Dermatol. 2014 Jul;39(5):583-9. doi: 10.1111/ced.12369. PMID 24934912
- [Result] Nofal A, Nofal E. Intralesional immunotherapy of common warts: successful treatment with mumps, measles and rubella vaccine. J Eur Acad Dermatol Venereol. 2010 Oct;24(10):1166-70. doi: 10.1111/j.1468-3083.2010.03611.x. PMID 20202055
- [Result] Jakhar D, Kaur I, Misri R. Intralesional vitamin D3 in periungual warts. J Am Acad Dermatol. 2019 May;80(5):e111-e112. doi: 10.1016/j.jaad.2018.11.007. Epub 2018 Nov 14. No abstract available. PMID 30447324
- [Result] Raghukumar S, Ravikumar BC, Vinay KN, Suresh MR, Aggarwal A, Yashovardhana DP. Intralesional Vitamin D3 Injection in the Treatment of Recalcitrant Warts: A Novel Proposition. J Cutan Med Surg. 2017 Jul/Aug;21(4):320-324. doi: 10.1177/1203475417704180. Epub 2017 Apr 6. PMID 28384048
- [Result] Aktas H, Ergin C, Demir B, Ekiz O. Intralesional Vitamin D Injection May Be an Effective Treatment Option for Warts. J Cutan Med Surg. 2016 Mar-Apr;20(2):118-22. doi: 10.1177/1203475415602841. Epub 2015 Aug 20. PMID 26294740
- [Result] Moscarelli L, Annunziata F, Mjeshtri A, Paudice N, Tsalouchos A, Zanazzi M, Bertoni E. Successful treatment of refractory wart with a topical activated vitamin d in a renal transplant recipient. Case Rep Transplant. 2011;2011:368623. doi: 10.1155/2011/368623. Epub 2012 Jan 3. PMID 23198256 (Retraction: PMID 35251733 Case Rep Transplant. 2022 Feb 23;2022:9838495)
- [Result] Raju J, Swamy A V, Swamy BLN, Raghavendra KR. INTRALESIONAL MEASLES , MUMPS AND RUBELLA ( MMR ) VACCINE-AN EFFECTIVE THERAPEUTIC TOOL IN THE TREATMENT OF WART . doi:10.18410/jebmh/2015/1176
- [Result] Chauhan PS, Mahajan VK, Mehta KS, Rawat R, Sharma V. The Efficacy and Safety of Intralesional Immunotherapy with Measles, Mumps, Rubella Virus Vaccine for the Treatment of Common Warts in Adults. Indian Dermatol Online J. 2019 Jan-Feb;10(1):19-26. doi: 10.4103/idoj.IDOJ_142_18. PMID 30775294
- [Result] El-Taweel AE, Salem RM, Allam AH. Cigarette smoking reduces the efficacy of intralesional vitamin D in the treatment of warts. Dermatol Ther. 2019 Mar;32(2):e12816. doi: 10.1111/dth.12816. Epub 2019 Jan 24. PMID 30623542
- [Result] Kavya M, Shashikumar BM, Harish MR, Shweta BP. Safety and Efficacy of Intralesional Vitamin D3 in Cutaneous Warts: An Open Uncontrolled Trial. J Cutan Aesthet Surg. 2017 Apr-Jun;10(2):90-94. doi: 10.4103/JCAS.JCAS_82_16. PMID 28852295
- [Result] Naseem R, Aamir S. The efficacy of intralesional measles, mumps, rubella (MMR) antigen in treatment of common warts. Pakistan J Med Heal Sci. 2013;7(4):1130-1133.
- [Result] Sobhy Mohamad N, Badran F, Yakout E. Evaluation of the efficacy of a combination - measles, mumps and rubella vaccine in the treatment of plantar warts. Our Dermatology Online. 2013;4(4):463-467. doi:10.7241/ourd.20134.118
- [Result] Shah A, Patel D, Ravishankar V. Measles, mumps and rubella vaccine as an intralesional immunotherapy in treatment of warts. Int J Res Med Sci. 2016;4(2):472-476. doi:10.18203/2320-6012.ijrms20160298
- [Result] Raju J, Swamy AV, Swamy BLN RK. Intralesional Measles, Mumps and Rubella (Mmr) Vaccine - an Effective Therapeutic Tool in the Treatment of Wart. J Evid Based Med Healthc. 2016;2(50):8548-8551. doi:10.18410/jebmh/2015/1176
- [Result] Rohit V, Gajula N. Role of Intralesional Measles Mumps Rubella Vaccine in Cutaneous Warts : A Case Control Study. 2017;(December):57-60.
- [Derived] Baaniya B, Marahatta S, Dahal R, Shah N. A Comparative Prospective Study to Assess Efficacy of Intralesional MMR (Measles, Mumps, Rubella) Vaccine and Intralesional Vitamin D3 in Treatment of Nongenital Warts. Health Sci Rep. 2025 May 5;8(5):e70782. doi: 10.1002/hsr2.70782. eCollection 2025 May. PMID 40330772

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Started | 33 | 33
Completed | 31 | 30
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3 | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.32 (11.167) | 23.93 (8.383) | 23.11 (9.847)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Brahmin/ Chhetri | 9 | 9 | 18
  Madhesi | 2 | 5 | 7
  Janajati | 18 | 14 | 32
  Others | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Nepal | 31 | 30 | 31
ITT population [Count of Participants; unit: Participants] | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of IL MMR and IL Vitamin D3 in Treatment of Warts
Description: Percentage of patients showing complete response to IL MMR and IL Vitamin D3
  Complete response -Complete disappearance of warts including distant ones and skin texture at the site is restored to normal (100%) Excellent response- Reduction in size and number including distant ones and few residual warts still visible (75-99%) Good response- Some reduction in size only including that of distant ones but no decrease in number of warts (50-74%) Poor or no response- No significant change in size and number of warts (0-49%)
Time Frame: Starting of treatment to end of three months follow-up after completing treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Participants
  Complete response | 25 | 22
  Excellent response | 2 | 6
  Good response | 3 | 1
  Poor or no response | 1 | 1

2. Secondary Outcome: Number of Participants in Each Education Level Group
Description: Distribution of wart patients into different education level like professional degree, graduate, intermediate, high school, middle school, primary school or illiterate
Time Frame: At the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Participants
  Graduate and higher | 2 | 4
  Intermediate | 4 | 2
  High School | 16 | 20
  Middle School | 6 | 3
  Primary and informal | 3 | 1

3. Secondary Outcome: Number of Participants in Each Occupation Group
Description: Number of participants with different occupations like professional, semiprofessional, clerical/shop/farm, skilled worker, semiskilled worker, unskilled worker, unemployed
Time Frame: At the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Participants
  Semiprofessional | 1 | 3
  Clerical/shop/farmer | 2 | 3
  Semiskilled | 1 | 4
  Unskilled | 1 | 1
  Unemployed | 3 | 1
  Student | 18 | 13
  Homemaker | 5 | 5

4. Secondary Outcome: Duration
Description: Duration of warts
Time Frame: At the time of enrollment
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
months | 24.2977 (23.99027) | 26.2417 (24.28020)

5. Secondary Outcome: Effect of the Warts on Patient's Life as Assessed by Dermatological Life Quality Index
Description: Quality of life (QoL) will be measured in wart patients, using the Nepali version of the dermatology life quality index (DLQI) questionnaire before initiation of treatment and at the end of follow up. DLQI contains 10 questions that involves 6 sections: symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Questions 1 and 2 assess symptoms and feelings; 3 and 4, daily activities; 5 and 6, leisure; 7, work and school; 8 and 9, personal relationships and 10, treatment.
  The DLQI consists of 10 questions. Each question is given 4 options from not at all effect (score 0) to very much effect (score 3). The minimum and maximum possible score, thus, is 0 and 30 respectively.
  Meaning of DLQI Scores 0-1 = no effect at all on patient's life 2-5 = small effect on patient's life 6-10 = moderate effect on patient's life 11-20 = very large effect on patient's life 21-30 = extremely large effect on patient's life
  .
Time Frame: At the time of enrollment and at the end of three months follow- up after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Participants
  no effect at all on patient's life | 9 | 10
  small effect on patient's life | 15 | 17
  moderate effect on patient's life | 6 | 1
  very large effect on patient's life | 1 | 2
  extremely large effect on patient's life | 0 | 0

6. Other Pre Specified Outcome: Number of Warts
Description: Number of warts in patients
Time Frame: At the time of enrollment
Measure: Mean (Standard Deviation); unit: Warts
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Warts | 21.58 (22.344) | 21 (31.107)

7. Other Pre Specified Outcome: Size
Description: Size range of warts
Time Frame: At the time of enrollment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
cm | 1.242 (0.9359) | 0.937 (0.5404)

8. Other Pre Specified Outcome: Number of Participants With Each Progression Type
Description: Number of participants with different progressions of warts like Gradual or rapid or stable or regressing lesions
Time Frame: At the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Participants
  Gradual | 23 | 27
  Rapid | 8 | 3

9. Other Pre Specified Outcome: Number of Participants Who Had Taken Past Treatment
Description: Frequency of different types of past treatment taken- either traditional or medical treatments
Time Frame: At the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
Number analyzed (Participants) | 31 | 30
Participants
  None | 21 | 19
  Traditional | 2 | 1
  Medical | 8 | 10

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Measles, Mumps, Rubella Vaccine | Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 6/30
Other Adverse Events (participants affected / at risk) | 31/31 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Measles, Mumps, Rubella Vaccine (N=31) | Vitamin D3 (N=30)
Hypervitaminosis D (Renal and urinary disorders) | 0 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Measles, Mumps, Rubella Vaccine (N=31) | Vitamin D3 (N=30)
Pain (Skin and subcutaneous tissue disorders) | 31 (31) | 30 (30)
Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT04428359/Prot_SAP_ICF_000.pdf